CLINICAL TRIAL: NCT01109771
Title: Absorbable Versus Permanent Mesh Fixation Trial in Laparoscopic Midline Ventral Hernia Repair (SORBET Trial)
Brief Title: Absorbable Versus Permanent Mesh Fixation Trial in Laparoscopic Midline Ventral Hernia Repair
Acronym: SORBET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/702
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Ventral Hernia
Keywords: Ventral hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- absorbable fixation left side (Active Comparator)
  Interventions: Device: permanent mesh fixation; Device: absorbable mesh fixation
- absorbable fixation right side (Active Comparator)
  Interventions: Device: permanent mesh fixation; Device: absorbable mesh fixation

INTERVENTIONS:
Device: permanent mesh fixation — Permanent mesh fixation will be used.
Device: absorbable mesh fixation — Absorbable mesh fixation will be used.

SUMMARY:
To compare the use of absorbable tackers versus permanent tack fixation using a polyester large pore mesh in laparoscopic midline ventral hernia repair in a multicenter (Belgian) prospective randomized single-blinded trial.

All patients referred for elective midline ventral hernia repair should be assessed for eligibility and entered in a study log, detailing all included patients during the study period.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from the adult patient (18 years and older, no maximum age)
* primary, incisional or recurrent midline ventral hernia requiring elective laparoscopic repair

Exclusion Criteria:

* no written informed consent
* hernia defects larger than 10cm diameter in width
* 'hostile' abdomen; open abdomen treatment
* contraindication to pneumoperitoneum
* emergency surgery (incarcerated hernia)
* lateral or parastomal hernia sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
number of patients with a VAS scale more than 40 | 1 year after surgery
  The Visual Analogue Scale (VAS) is commonly used to measure the intensity of pain or other subjective experiences. It is a simple and effective tool.
  The VAS consists of a straight line, usually 10 cm long, with endpoints defining extreme limits such as 'No pain' and 'Worst imaginable pain'. Respondents mark a point on the line that represents their perception of their current state.
  Scoring:
  Scale Title: Visual Analogue Scale (VAS) Minimum Value: 0 (indicating no pain or the least possible experience of the measured parameter) Maximum Value: 10 (indicating worst imaginable pain or the most extreme experience of the measured parameter) Higher Scores: Indicate a worse outcome (e.g., more intense pain or greater severity of the measured parameter).

SECONDARY OUTCOMES:
number of invasive interventions (local infiltrations, reoperations) postoperatively | 1 year after surgery
  number of invasive interventions (local infiltrations, reoperations) postoperatively, 1 year after surgery
number of patients taking analgetics using MCGill painscore | 1 year post-surgery
  The McGill Pain Questionnaire (MPQ) measures the quality and intensity of pain through three components:
  Pain Rating Index (PRI): Derived from 78 pain descriptors in four categories: Sensory (S), Affective (A), Evaluative (E), Miscellaneous (M). Each descriptor has a numerical value.
  Scale Title: Pain Rating Index (PRI) Range: 0-78 Higher Scores: Indicate greater intensity of pain. Present Pain Intensity (PPI): A single-item scale rating current pain on a 6-point scale.
  Scale Title: Present Pain Intensity (PPI) Range: 0 (No Pain) to 5 (Excruciating Pain) Higher Scores: Indicate greater intensity of pain. Number of Words Chosen (NWC): Total pain descriptors selected. Scale Title: Number of Words Chosen (NWC) Range: 0-20 Higher Scores: Indicate more complex or severe pain.
perioperative morbidity rate | 1 year after surgery
  perioperative morbidity rate, 1 year after surgery
quality of life by using EQ5D score | 1 year post-surgery
  The EQ-5D is a standardized instrument for measuring generic health status, providing a descriptive profile and a single index value.
  Descriptive System: Comprises five dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression. Each dimension has three severity levels: No problems, Some problems, Extreme problems. Responses form a five-digit number describing the health state (e.g., 11223).
  EQ Visual Analogue Scale (EQ VAS): Records self-rated health on a vertical scale from 0 (Worst health) to 100 (Best health), quantifying the patient's overall health perception.
  EQ-5D Index Value: Derived from the descriptive system. Scale Title: EQ-5D Index Value Range: Typically -0.594 to 1 Higher Scores: Indicate better health outcomes.
recurrence rate | 1 year post-surgery
  recurrence rate, 1 year post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, Principal Investigator — University Hospital, Ghent
Locations (11):
- Belgium (11):
  - Virga Jesseziekenhuis, Hasselt, Limburg
  - Imelda Ziekenhuis, Bonheiden
  - CHU Charleroi, Charleroi
  - St-Vincentius Ziekenhuis, Deinze
  - AZ Sint-Dymphna, Geel
  - University Hospital Ghent, Ghent
  - Ziekenhuis Maas en Kempen, Maaseik
  - AZ Sint-Maarten, Mechelen
  - Heilig Hart Ziekenhuis, Mol
  - UCL Mont-Godinne, Namur
  - H. Serruys Ziekenhuis, Ostend

REFERENCES:
- See also: website University Hospital Ghent — http://www.uzgent.be